CLINICAL TRIAL: NCT05682872
Title: Multifactorial Fall Prevention Program in People Aged 65 or Over of an Urban Area of Talavera de la Reina
Brief Title: Multifactorial Fall Prevention Program
Acronym: Dodgers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Castilla-La Mancha Health Service (Other)
Collaborators: Colegio Oficial de Terapeutas Ocupacionales de Castilla - La Mancha (Unknown); Fundación Eurocaja Rural (Unknown); Fundación Hestia (Unknown); Unidad de Apoyo a la Investigación de la Gerencia de Atención Integrada de Talavera de la Reina (Unknown); Decathlon España S.A.U. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 57/2020
Record Dates: First submitted 2022-12-13; First posted 2023-01-12 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Frail Elderly Syndrome
Keywords: risk of falls; prevention; clinical trial

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Experimental group receive multifactorial intervention (based on the GBPC "Prevention of Falls and reduction of Injuries derived from falls" - RNAO).
  Interventions: Behavioral: Physical exercise program (VIVIFRAIL) supervised by a physiotherapist; Behavioral: Adequacy of the environment; Behavioral: Polypharmacy review; Behavioral: Health education related to falls prevention (4 sessions); Behavioral: General Assement; Behavioral: Evaluation of patients by an expert group; Behavioral: Information brochures on the importance of physical exercise
- Control Group (Active Comparator): Control group receive activities on falls prevention by Primary Care professionals on a care routine.
  Interventions: Behavioral: Information brochures on the importance of physical exercise; Behavioral: Physical exercise program (VIVIFRAIL) supervised by a primary care doctor or primary care nurse; Behavioral: Regular assessment and follow-up by primary care doctor and primary care nurse; Behavioral: Health education related to falls prevention (1 session)

INTERVENTIONS:
Behavioral: Physical exercise program (VIVIFRAIL) supervised by a physiotherapist — Promotion of physical exercise program for frailty and falls prevention in elderly. Muscular strength training, cardiovascular resistance, balance and gait. Initially guided and supervised every 3 months by a physiotherapist.
  Arms: Experimental Group
Behavioral: Adequacy of the environment — A home study and the environment will be made to diagnose fall risks. Guided and supervised by a occupational therapist during a home visit.
  Arms: Experimental Group
Behavioral: Polypharmacy review — Assessment of the medication that patients receives related to fall risks proposing its adjustment. Revised by a primary care doctor different from care routine.
  Arms: Experimental Group
Behavioral: Health education related to falls prevention (4 sessions) — SESSION 1: Fall Risk factors. Pharmacology. Nutrition and falls (Primary Care Doctor and Primary Care Nurse)
  SESSION 2: Accident prevention through environmental modification (Occupational Therapist)
  SESSION 3: Importance of physical exercise to prevent falls (Physiotherapist)
  SESSION 4: Footwear and foot care. How to react to a fall?: what to do and how to get up? (Primary Care Nurse)
  Arms: Experimental Group
Behavioral: General Assement — General assessment (feet, footwear, nutrition, cognitive/psychological, social of risk factors) carried out by Primary Care Doctor and Primary Care Nurse
  Arms: Experimental Group
Behavioral: Evaluation of patients by an expert group — Evaluation of the patient by an expert group (Primary care doctor, primary care nurse, polypharmacy review doctor, occupational therapist, frailty group) and decision-making for correction of fall risk factors.
  Arms: Experimental Group
Behavioral: Information brochures on the importance of physical exercise — Integrated Assistance Process for prevention falls in elderly. Benefits of physical exercise and fall prevention at home. Prepared by the Junta de Comunidades de Castilla-La Mancha and Servicio de Salud de Castilla-La Mancha.
Behavioral: Physical exercise program (VIVIFRAIL) supervised by a primary care doctor or primary care nurse — Promotion of physical exercise program for frailty and falls prevention in elderly. Muscular strength training, cardiovascular resistance, balance and gait. Supervised by primary care doctor o primary care nurse according to passport recommendations.
  Arms: Control Group
Behavioral: Regular assessment and follow-up by primary care doctor and primary care nurse — General assessment related to falls with the established protocols at primary care routine.
  Arms: Control Group
Behavioral: Health education related to falls prevention (1 session) — There will be a single session. The session will cover the following topics: Fall Risk factors. Pharmacology. Nutrition and falls. Accident prevention through environmental modification. Importance of physical exercise to prevent falls. Footwear and foot care. How to react to a fall?: what to do and how to get up?
  Arms: Control Group

SUMMARY:
The main objective is evaluate the effectiveness of a Multifactorial Pilot Program on the Prevention of Falls in people aged 65 or over during 4 years at Gerencia de Atención Integrada de Talavera de la Reina.

DETAILED DESCRIPTION:
Introduction: Falls are a major global public health problem. Falls are the second leading cause of death from unintentional injuries in the world. The highest mortality rates correspond to 60 years old people. 20-30% suffer from moderate-serious injuries (hip fractures, head injuries...), that reduce mobility and independence, increasing the risk of premature death. Moreover, there are more than 400 risk factors. Most can be modified to decrease the risk of falling.

Objective: To evaluate the effectiveness of a Multifactorial Pilot Program on the Prevention of Falls in people aged 65 or over during 4 years at Gerencia de Atención Integrada de Talavera de la Reina.

Material and methods: Randomized clinical trial with 264 patients is carried out. 65 years old or older patients are recruited from primary care (≥ 1 positive response in the Frailty Screening Test, or ≥ 3 in the Downton Test and > 90 in the Barthel Index). Falls risk is assessed using validated scales. Experimental group receive multifactorial intervention (based on the GBPC "Prevention of Falls and reduction of Injuries derived from falls" - RNAO). Control group receive recommendations (physical exercise, health education on risk factors, footwear, exercise, home adaptation, nutrition, …). Variables are presented with their frequency distribution. Qualitative variables as median and range, and quantitatives with their mean and standard deviation. Association between qualitative variables are evaluated with Pearson's Chi-square test. Student's t test be used when the distribution of the variable adjusts to normality. The null hypothesis will be rejected with an error α less than 0.05.

Expected benefits: It is expected to reduce the risk of falls in 30-35% of 65 years old people or older in the urban area of Talavera de la Reina. It would mean great savings and improve the quality of life. It is expected to increase the years of healthy life. It is intended to provide health professionals with a tool to make clinical decisions based on evidence on the prevention of falls to be used as a unified work protocol at Gerencia de Atención Integrada de Talavera de la Reina.

ELIGIBILITY:
Inclusion Criteria:

* 65 years old or older patients
* Live in Talavera de la Reina
* Ability to walk at the Health Center
* ≥ 3 in the Downton Test
* > 90 in the Barthel Index
* Sign the informed consent

Exclusion Criteria:

* Patients with an intense physical activity
* Use of a wheelchair
* Amputations or prosthetic limbs
* Deafness
* Blindness
* Moderate or severe cognitive impairment
* Vertebral, pelvic or lower limb fractures in the 12 months prior to entering the program
* Absolute contraindication to physical exercise

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2021-03-09 (Actual); Primary Completion 2026-10-09 (Estimated); Study Completion 2026-11-09 (Estimated)

PRIMARY OUTCOMES:
Number of falls | 24 months after intervention
  To assess the number of falls in the intervention group and control group to determine if the intervention group has a significantly lower rate of falls.

SECONDARY OUTCOMES:
Number of falls that have been treated in hospital | 24 months after intervention
  Evaluate the number of falls that have been treated in hospital due to fractures or trauma resulting from falls
Euroqol-5D-5L | 24 months after intervention
  Evaluate the impact on the quality of life in people over 65 years of age who live in the community and who participate in this program

CONTACTS AND LOCATIONS:
Overall Officials: Nuria García Bonilla, Principal Investigator — Gerencia de Atención Integrada de Talavera de la Reina
Locations (1):
- Gerencia de Atención Integrada de Talavera de la Reina, Talavera de la Reina, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aranda-Gallardo M, Morales-Asencio JM, Canca-Sanchez JC, Toribio-Montero JC. Circumstances and causes of falls by patients at a Spanish acute care hospital. J Eval Clin Pract. 2014 Oct;20(5):631-7. doi: 10.1111/jep.12187. Epub 2014 Jun 5. PMID 24902772
- [Background] Viana TS, Martin MR, Crespo FN, Rodriguez EM, Merino GM, Ruiz JM, Lorenzo IL, Quintas CG. [What is the real incidence of falls in hospitals?]. Enferm Clin. 2011 Sep-Oct;21(5):271-4. doi: 10.1016/j.enfcli.2011.02.011. Epub 2011 Jun 30. Spanish. PMID 21719335
- [Background] Silva Gama ZA, Gomez Conesa A, Sobral Ferreira M. [Epidemiology of falls in the elderly in Spain: a systematic review, 2007]. Rev Esp Salud Publica. 2008 Jan-Feb;82(1):43-55. doi: 10.1590/s1135-57272008000100004. Spanish. PMID 18398550
- [Background] Ambrose AF, Cruz L, Paul G. Falls and Fractures: A systematic approach to screening and prevention. Maturitas. 2015 Sep;82(1):85-93. doi: 10.1016/j.maturitas.2015.06.035. Epub 2015 Jun 26. PMID 26255681
- [Background] Gillespie LD, Robertson MC, Gillespie WJ, Sherrington C, Gates S, Clemson LM, Lamb SE. Interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2012 Sep 12;2012(9):CD007146. doi: 10.1002/14651858.CD007146.pub3. PMID 22972103
- [Background] Hopewell S, Adedire O, Copsey BJ, Boniface GJ, Sherrington C, Clemson L, Close JC, Lamb SE. Multifactorial and multiple component interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2018 Jul 23;7(7):CD012221. doi: 10.1002/14651858.CD012221.pub2. PMID 30035305
- [Background] Sherrington C, Michaleff ZA, Fairhall N, Paul SS, Tiedemann A, Whitney J, Cumming RG, Herbert RD, Close JCT, Lord SR. Exercise to prevent falls in older adults: an updated systematic review and meta-analysis. Br J Sports Med. 2017 Dec;51(24):1750-1758. doi: 10.1136/bjsports-2016-096547. Epub 2016 Oct 4. PMID 27707740
- [Background] Kyrdalen IL, Moen K, Roysland AS, Helbostad JL. The Otago Exercise Program performed as group training versus home training in fall-prone older people: a randomized controlled Trial. Physiother Res Int. 2014 Jun;19(2):108-16. doi: 10.1002/pri.1571. Epub 2013 Dec 11. PMID 24339273
- [Background] Izquierdo M, Casas-Herrero A, Zambm-Ferraresi F, Martínez-Velilla N, Alonso-Bouzón C, Rodríguez-Mañas L, et al. A Practical Guide for Prescribing a Multi-Component Physical Training Program to prevent weakness and falls in People over 70. 2017. http://www.vivifrail.com/resources.
- [Background] Sepulveda-Loyola W, Rodriguez-Sanchez I, Perez-Rodriguez P, Ganz F, Torralba R, Oliveira DV, Rodriguez-Manas L. Impact of Social Isolation Due to COVID-19 on Health in Older People: Mental and Physical Effects and Recommendations. J Nutr Health Aging. 2020;24(9):938-947. doi: 10.1007/s12603-020-1469-2. PMID 33155618
- [Background] Jutkowitz E, Gitlin LN, Pizzi LT, Lee E, Dennis MP. Cost effectiveness of a home-based intervention that helps functionally vulnerable older adults age in place at home. J Aging Res. 2012;2012:680265. doi: 10.1155/2012/680265. Epub 2011 Aug 16. PMID 21876812
- See also: World Health Organization. falls. Fact Sheet no 344. — http://www.who.int/mediacentre/factsheets/fs344/es/
- See also: A CDC Compendium of Effective Fall Interventions: What Works for Community-Dwelling Older Adults — https://www.cdc.gov/falls/pdf/cdc_falls_compendium-2015-a.pdf